CLINICAL TRIAL: NCT05968352
Title: Restoration of Bladder Function in Spinal Cord Injury
Status: Withdrawn | Type: Observational
Why Stopped: Unable to find participants to recruit
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS 260021
Record Dates: First submitted 2023-07-20; First posted 2023-08-01 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-10

CONDITIONS: Bladder Dysfunction; Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Sacral Anterior Root Stimulation (SARS) — Comparison of High frequency versus low frequency stimulation

SUMMARY:
The aim of this study is to develop improved methods of restoring function to the neurogenic bladder, using electrical stimulation without cutting nerves in patients with spinal cord injury.

The investigators will test 5-10 subjects with existing sacral anterior root stimulation (SARS) devices and look at the effects of high frequency (up to 600Hz) compared to the usual low frequency stimulation on bladder function. The investigators are particularly interested in whether it is possible to reproduce a 'functional' dorzal rhizotomy using high frequency stimulation of the S2 efferent nerves

DETAILED DESCRIPTION:
This is a proof of concept study of the effects on the urinary bladder and sphincter of high frequency stimuli applied to sacral efferent nerves. The effects on the bladder of low frequency stimuli applied to sacral afferent nerves will also be studied. It is also part of an academic collaboration between Oxford and Stanford University. The results will not be sold to Stanford but will be shared to enhance the development of therapies for patients with spinal cord injury. There is no intention to commercialise the findings at this stage nor to use the data for CE-marking.

Participants will be patients with clinically complete spinal cord injury who already have a commercially available implanted Finetech Brindley bladder stimulator with electrodes on the sacral nerves or roots, controlled by an external transmitter whose frequency can be adjusted by the investigator. This study will explore modified stimulation parameters and will deliver the stimulation pattern with a modified/experimental external stimulation control unit. The motivation for exploring these parameters is to see if clinical efficacy might be improved for future systems.

Primary outcome: Measurement of the effects of high and low frequency stimulation of the sacral efferent nerves on Bladder Pressure, rectal pressure, Detrusor pressure, Sphincter pressure, volume voided, post-void residual volume, voiding flow rate

Secondary measures: Effects of low frequency stimulation on bladder pressure, bladder capacity and reflex incontinence

The exploration of these novel stimulation parameters will require modification of the existing CE-marked system. The modifications will be limited to the external stimulation control unit, and will not compromise either the implantable system or its capability to continue normal operation with the existing CE-marked external control unit. The modified external stimulation control unit will be referred to as the "research stimulation controller." The use environment for the research stimulation controller will be a controlled hospital/laboratory setting, under clinical supervision. Outside of the clinic, the CE-marked system will be used to ensure normal therapy is provided to the subject. Access to the research stimulation controller will be controlled by the PI to prevent inadvertent misuse.

The development of the research stimulation controller will follow accepted good design practices. More specifically, the team will use a scaled version of 13845-compliant processes to 1) assess user needs 2) generate a risk analysis and plan 3) develop system requirements from design inputs 4) document and summarize design outputs 5) perform device verification tests and 6) perform user validation tests. These files will be maintained in a controlled document system.

The modified controller is similar to the CE marked device but will allow the investigators to explore a wider range of electrical stimulation parameters such as different waveforms and higher frequencies. Our intention is to use up to 600 Hz frequencies, compared to the existing frequencies in this device of up to 53 Hz. These changes are modest and are well within the energy delivery provided by existing commercial neuromodulation systems such as spinal cord stimulation (typical parameters for spinal cord stimulation include the Nevro® system that delivers up to 10kHz). Patients both with and without posterior sacral rhizotomy will also be included. No further surgery is required. Measurements of bladder function will be made in the urodynamic laboratory.

The study is prospective and unblinded. Each participant will serve as their own control; outcome measures will be compared with different frequencies of electrical stimuli and with no electrical stimuli.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinically complete spinal cord injury who have undergone implantation of a Finetech Brindley Bladder controller, with or without sacral posterior rhizotomy.
* Male or female, aged 18 years or over.
* Patients willing and able to give informed consent to involvement in the study

Exclusion Criteria:

* External urethral sphincterotomy
* Patients are taking part in any studies on drugs or devices that alter bladder or autonomic function
* Any other significant comorbidity or illness that would preclude their participation or increase the risk to them of participating in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with clinically complete spinal cord injury who have undergone implantation of a Finetech Brindley Bladder Controller, with or without sacral posterior rhizotomy. John Radcliffe Hospital (Oxford), Royal National Orthopaedic Hospital (Stanmore) and Walton Centre (Liverpool) will be both patient identification centres and research sites for this study. Stoke Mandeville Hospital will be an additional patient identification centre, but studies on patients identified there will be conducted at Oxford as patients are generally under joint care between Stoke Mandeville Hospital and Oxford.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-11-18 (Actual); Primary Completion 2025-10-14 (Actual); Study Completion 2025-10-14 (Actual)

PRIMARY OUTCOMES:
Bladder Pressure | 2-3 hours
  Urodynamics testing - High frequency SARS
Rectal Pressure | 2-3 hours
  Urodynamics- High frequency SARS
Detrusor Pressure | 2-3 hours
  Urodynamics- High frequency SARS
Sphincter Pressure | 2-3 hours
  Urodynamics1- High frequency SARS
Volume voided | 2-3 hours
  urodynamics- High frequency SARS
Post-void residual volume | 2-3 hours
  Urodynamics- High frequency SARS
Voiding Flow Rate | 2-3 hours
  Urodynamics- High frequency SARS

SECONDARY OUTCOMES:
Bladder pressure | 2-3 hours
  Urodynamics - Low frequency SARS
Bladder Capacity | 2-3 hours
  Urodynamics - Low frequency SARS
Reflex incontinence | 2-3 hours
  Urodynamics - Low frequency SARS

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oxford, Oxford, Oxon, United Kingdom

IPD SHARING:
Plan to Share IPD: No